CLINICAL TRIAL: NCT03153813
Title: Efficacy And Safety Of High Concentration Capsaicin Patches In Knee Osteoarthritis In Obese Patients: A Randomized Prospective Double Blind Placebo Controlled Study
Brief Title: Capsaicin Patches In Knee Osteoarthritis In Obese Patients
Acronym: CHILI-OB
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Nadine ATTAL (Other)
Responsible Party: Sponsor-Investigator, Nadine ATTAL, Co-investigator, Hospital Ambroise Paré Paris
Organization: Hospital Ambroise Paré Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CHILI-OB
Record Dates: First submitted 2015-11-04; First posted 2017-05-15 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Pain
Keywords: pain; knee osteoarthritis; obesity; capsaicin
MeSH Terms: conditions — Pain; Osteoarthritis, Knee; Obesity | interventions — Capsaicin; Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug (Experimental): Up to 4 patches to cover a surface of 1200 cm2 will be applied to the painful area depending on the surface of pain during 60 minutes : capsaicin 8% patches (Qutenza)
  Interventions: Drug: capsaicin 8% patches (Qutenza)
- Placebo (Placebo Comparator): Up to 4 patches will be applied to the painful area depending on the surface of pain during 60 minutes : placebo
  Interventions: Other: Placebo patches

INTERVENTIONS:
Drug: capsaicin 8% patches (Qutenza)
  Arms: Drug
Other: Placebo patches
  Arms: Placebo

SUMMARY:
To assess the efficacy and safety of high concentration capsaicin patches in pain due to osteoarthritis (OA) of the knee in patients with obesity

DETAILED DESCRIPTION:
Osteoarthritis is one of the leading causes of pain and disability. In France osteoarthritis of the knee, the most common form of osteoarthritis has been recently estimated to affect 4.7 % of men and 2.5 % of women .

One particularly exposed population to osteoarthritis is represented by obese patients. Obesity, defined as a body mass index (BMI) above 30 kg/m², is considered to be one of the most important risk factors for osteoarthritis (OA) in knees. Numerous longitudinal studies show a strong association between obesity, and radiographic knee OA, e.g. in the Framingham Study, the Chingford Study, the Baltimore Longitudinal Study of Aging, the John Hopkins Precursors Study, and in longitudinal studies in UK and the Netherlands. Thus, the WHO initiative on counteracting obesity also accepts OA as a consequence of obesity . Each BMI increase by 1 kg/m² is associated with a 15% increased risk of OA. A number of recent studies involving the association between obesity and knee osteoarthritis have since been published. A large, population-based prospective study (n = 823) conducted by Toivanen et al. with a follow-up of 22 years found that the risk for knee osteoarthritis was 7 times greater for people with BMI ≥30 compared to the control of people with BMI <25. A prospective cohort study of the Norwegian population by Grotle et al. (10) that followed 1,675 patients reported that BMI >30 was significantly associated with osteoarthritis of the knee, with odds ratio of 2.81, and 95% CI of 1.32-5.96. Lohmander et al. found that in a large cohort study of 27,960 patients from the Swedish population, the relative risk for knee osteoarthritis (fourth quartile compared to first quartile) was 8.1, with a 95% CI of 5.3-12.4. Finally, a case-control study from Holliday et al. with 1,042 knee osteoarthritis patients and 1,121 matched controls reported that the adjusted odds ratio for knee osteoarthritis in patients with BMI >30 was 7.48 with 95% CI of 5.45-10.27.

Pain is one of the major comorbid conditions that may preclude effective weight management in these patients, particularly with regards to physical activity, since pain increases with effort and movement. Obese patients generally receive oral analgesics, such as weak opioids or tramadol, but due to a number of associated comorbidities, they generally do not tolerate, or have contraindications to, centrally acting analgesics. Furthermore an increasing number of obese patients are managed by malabsorbtive bariatric surgical procedures, exposing them at risk for inefficacity by oral analgesics, in regards to the malabsorptive effect.

Therefore alternative therapies, and in particular topical treatments, may be indicated in these patients as these drugs have less systemic side effects. The use of such treatments in patients with obesity should contribute to facilitate rehabilitation and hence contribute to weight loss, which may further help to reduce pain.

One promising topical treatment is represented by capsaicin. Capsaicin is an agonist of the transient receptor potential vanilloid 1 (TRPV1), a non-selective cation channel. It is well established that capsaicin applied in high concentration to the skin can cause initial nociceptor sensitization through its agonistic effects on TRPV1 receptors then subsequently acts in the skin to attenuate cutaneous hypersensitivity and reduce pain by a process best described as "defunctionalisation" of nociceptor fibres (e.g. temporary loss of membrane potential, inability to transport neurotrophic factors leading to altered phenotype, and reversible retraction of epidermal and dermal nerve fibre terminals). Evidence suggests that the utility of topical capsaicin may extend beyond painful peripheral neuropathies, and that this treatment may be particularly relevant in patients with osteoarthritis pain. Thus TRPV1 is mainly expressed by nociceptive neurons in dorsal root and trigeminal ganglia. However, there is increasing evidence that TRPV1 is also expressed in various cell types including synovial fibroblasts (SF) from patients with symptomatic osteoarthritis (OA) and thus may play a role in non-neuronal mechanisms that might modulate nociception in symptomatic osteoarthritis.

An additional effect of high concentration of capsaicin, which does not involve TRPV1, is a direct inhibition of mitochondrial respiration. Furthermore, by using the approach of patch-clamp, capsaicinoids (capsaicin and dihydrocapsaicin) have been shown to reversibly inhibit the currents of T-type voltage-dependent Ca2+channels, suggesting the effect of capsaicinoids on pain relief may also be related to the inhibition of T-type Ca2+ channels.

Capsaicin is metabolized rapidly by several cytochrome enzymes present in human liver, but in vitro studies shows that its metabolism in human skin is quite low. Capsaicin reside at the site of action (i.e. skin) relatively unchanged, whereas capsaicin which is transdermally absorbed is rapidly eliminated and does not have any systemic effect.

To date, repeated applications of low dose capsaicin cream at different concentrations (0.0125 to 0.25 %) have been found moderately effective in OA of the knee or hand, based on the basis of six double or single blind trials with sample sizes ranging from 14 to 200 patients. However repeated applications of capsaicin cream are difficult on the long term particularly because of the burning sensation induced by the cream and the necessity to repeat applications several times per day.

Recently high concentration capsaicin patches (8%) (Qutenza) have been developed for the treatment of peripheral neuropathic pain. These treatments induce long lasting analgesic effects in these conditions lasting up to an average of 3 months after a 30 to 60 minutes application. The burning side effect related to the application of the patch is rapidly reversible and very few severe side effects have been reported with this procedure.

If the primary cause of chronic musculoskeletal pain lies deep within joints and topical capsaicin does not provide substantial transdermal delivery, then the apparent efficacy of topical capsaicin in lower back pain and OA could be postulated to be by CNS modulatory mechanisms. Another possibility is that alterations in, or sensitization of, cutaneous nociceptors could be a contributing factor. Such alterations might be driven by unusually high concentrations of cytokines or growth factors in joints which could either diffuse some distance away from the primary site of inflammation or promote excitatory phenotypes in nearby collateral axons. Furthermore there is increasing evidence that TRPV1 expression is not limited to primary afferent neurons but that the receptor is expressed in various cell types throughout the body. TRPV1 is present in synovial fibroblasts from symptomatic OA and RA (rheumatoid arthritis) patients and the receptor can be activated by stimulation with the vanilloid capsaicin. It is very likely that capsaicin stimulation does not only induce IL-6 production but also results in the release of other signalling molecules that may transfer the information to other non-neuronal or neuronal cells and thereby contribute to a modulation of nociception in the inflamed joint.

Based on the mechanisms described above, there are reasons to believe that Qutenza may also be effective in osteoarthritis pain. To date, there are strictly no data regarding potential efficacy and safety of this treatment in osteoarthritis pain in obese patients

ELIGIBILITY:
Inclusion Criteria:

* Enrolled patients will be males or females,
* aged over 18 years,
* have pain for at least 3 months due to mild to moderate osteoarthritis of the knee (meeting American College of Rheumatology clinical and radiographic criteria), of at least moderate intensity (pain intensity score over the last 24 hours before enrolment ≥ 4/10),
* with a BMI above 30 kg/m²
* and no other pain conditions accounting for their disability.
* The skin will be intact and no blessed.
* All female patients should take contraception during all study and at least 30 days after closer.
* All patients must sign informed consent.
* All patients will be recruited from the Department of Nutrition, Ambroise Paré University Hospital and treatment will be given during a dedicated day care clinic.

Exclusion Criteria:

* Patients necessitating surgery,
* with relative contraindications to capsaicin patches, particularly with unstable hypertension or cardiac condition,
* past history of capsaicin use will not be included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-07; Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Effects on self reported average pain intensity on pain diaries throughout the study (on NRS from 0 to 10) | Over the 3 months of the study
  The primary outcome measure will be the reduction of average pain intensity as assessed by the patients daily using a pain diary throughout the 3 months of the study. The comparison will be made with baseline pain values started 7 days before the treatment.

SECONDARY OUTCOMES:
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain, function and stiffness | at each follow up period 1, 2 and 3 months as compared to baseline values
  WOMAC pain and function index
safety as assessed by side effects during and after application | during and immeditaly after application and at each follow up period 1, 2 and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Claire Carette, Principal Investigator — Hospital Ambroise Pare Paris
Locations (1):
- Hospital Ambroise Paré, Nutrition Department, Boulogne-Billancourt, France